CLINICAL TRIAL: NCT01226784
Title: The Effects of Training and Relaxation on Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Sahlgrenska University Hospital (Other); University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Eva Kosek, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RF 2010 stud GLS
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
Keywords: Strength exercise; Physical exercise; Physiotheraphy
MeSH Terms: conditions — Fibromyalgia; Motor Activity

ARMS (2):
- Physcial exercise (Active Comparator): 15 weeks of progressive resistance group exercise, twice/week supervised by physical therapist
  Interventions: Behavioral: Physcial activity
- Relaxation exercise (Active Comparator): 15 weeks of relaxation exercise, twice/week supervised by physical therapist
  Interventions: Behavioral: Physcial activity

INTERVENTIONS:
Behavioral: Physcial activity — Strenght training Relaxation exercise

SUMMARY:
Effects of physical training and relaxation exercise on pathophysiological mechanisms and symptoms in finbromyalgia patients.

DETAILED DESCRIPTION:
A multi-center trial examining the effects of progressive resistance group exercise compared with an active control group (relaxation). A person-centred model of exercise was used. The intervention was performed twice a week for 15 weeks and was supervised by experienced physiotherapists.

Secondary aims off this multi-center study was to improve the understanding of pain mechanisms in fibromyalgia and how these are affected by physical exercise. Please see references of published articles for details.

ELIGIBILITY:
Inclusion Criteria: ACR 1990 criteria for fibromyalgia -

Exclusion Criteria: Other dominating pain condition, severe disease preventing from participating in physical exercise

-

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Muscle function | 2010-2013
  isometric knee-extension force (Steve Strong®)

SECONDARY OUTCOMES:
Fibromyalgia impact questionnaire | 2010-2013
  Ratings on FIQ, total score
VAS pain | 2010-2013
  Pain intensity ratings on VAS

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Linkopings University Hospital, Linköping
  - Karolinska Institute, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahlen K, Ernberg M, Kosek E, Mannerkorpi K, Gerdle B, Ghafouri B. Significant correlation between plasma proteome profile and pain intensity, sensitivity, and psychological distress in women with fibromyalgia. Sci Rep. 2020 Jul 27;10(1):12508. doi: 10.1038/s41598-020-69422-z. PMID 32719459
- [Background] Stensson N, Gerdle B, Ernberg M, Mannerkorpi K, Kosek E, Ghafouri B. Increased Anandamide and Decreased Pain and Depression after Exercise in Fibromyalgia. Med Sci Sports Exerc. 2020 Jul;52(7):1617-1628. doi: 10.1249/MSS.0000000000002293. PMID 32168104
- [Background] Jablochkova A, Backryd E, Kosek E, Mannerkorpi K, Ernberg M, Gerdle B, Ghafouri B. Unaltered low nerve growth factor and high brain-derived neurotrophic factor levels in plasma from patients with fibromyalgia after a 15-week progressive resistance exercise. J Rehabil Med. 2019 Oct 29;51(10):779-787. doi: 10.2340/16501977-2593. PMID 31544950
- [Background] Stensson N, Ghafouri N, Ernberg M, Mannerkorpi K, Kosek E, Gerdle B, Ghafouri B. The Relationship of Endocannabinoidome Lipid Mediators With Pain and Psychological Stress in Women With Fibromyalgia: A Case-Control Study. J Pain. 2018 Nov;19(11):1318-1328. doi: 10.1016/j.jpain.2018.05.008. Epub 2018 Jun 7. PMID 29885369
- [Background] Larsson A, Palstam A, Bjersing J, Lofgren M, Ernberg M, Kosek E, Gerdle B, Mannerkorpi K. Controlled, cross-sectional, multi-center study of physical capacity and associated factors in women with fibromyalgia. BMC Musculoskelet Disord. 2018 Apr 19;19(1):121. doi: 10.1186/s12891-018-2047-1. PMID 29673356
- [Background] Ernberg M, Christidis N, Ghafouri B, Bileviciute-Ljungar I, Lofgren M, Bjersing J, Palstam A, Larsson A, Mannerkorpi K, Gerdle B, Kosek E. Plasma Cytokine Levels in Fibromyalgia and Their Response to 15 Weeks of Progressive Resistance Exercise or Relaxation Therapy. Mediators Inflamm. 2018 Apr 18;2018:3985154. doi: 10.1155/2018/3985154. eCollection 2018. PMID 29849487
- [Background] Larsson A, Palstam A, Lofgren M, Ernberg M, Bjersing J, Bileviciute-Ljungar I, Gerdle B, Kosek E, Mannerkorpi K. Pain and fear avoidance partially mediate change in muscle strength during resistance exercise in women with fibromyalgia. J Rehabil Med. 2017 Nov 21;49(9):744-750. doi: 10.2340/16501977-2278. PMID 29068036
- [Background] Tour J, Lofgren M, Mannerkorpi K, Gerdle B, Larsson A, Palstam A, Bileviciute-Ljungar I, Bjersing J, Martin I, Ernberg M, Schalling M, Kosek E. Gene-to-gene interactions regulate endogenous pain modulation in fibromyalgia patients and healthy controls-antagonistic effects between opioid and serotonin-related genes. Pain. 2017 Jul;158(7):1194-1203. doi: 10.1097/j.pain.0000000000000896. PMID 28282362
- [Background] Martinsen S, Flodin P, Berrebi J, Lofgren M, Bileviciute-Ljungar I, Mannerkorpi K, Ingvar M, Fransson P, Kosek E. The role of long-term physical exercise on performance and brain activation during the Stroop colour word task in fibromyalgia patients. Clin Physiol Funct Imaging. 2018 May;38(3):508-516. doi: 10.1111/cpf.12449. Epub 2017 Jun 18. PMID 28627125
- [Background] Bjersing JL, Larsson A, Palstam A, Ernberg M, Bileviciute-Ljungar I, Lofgren M, Gerdle B, Kosek E, Mannerkorpi K. Benefits of resistance exercise in lean women with fibromyalgia: involvement of IGF-1 and leptin. BMC Musculoskelet Disord. 2017 Mar 14;18(1):106. doi: 10.1186/s12891-017-1477-5. PMID 28288611
- [Background] Gerdle B, Ernberg M, Mannerkorpi K, Larsson B, Kosek E, Christidis N, Ghafouri B. Increased Interstitial Concentrations of Glutamate and Pyruvate in Vastus Lateralis of Women with Fibromyalgia Syndrome Are Normalized after an Exercise Intervention - A Case-Control Study. PLoS One. 2016 Oct 3;11(10):e0162010. doi: 10.1371/journal.pone.0162010. eCollection 2016. PMID 27695113
- [Background] Ericsson A, Palstam A, Larsson A, Lofgren M, Bileviciute-Ljungar I, Bjersing J, Gerdle B, Kosek E, Mannerkorpi K. Resistance exercise improves physical fatigue in women with fibromyalgia: a randomized controlled trial. Arthritis Res Ther. 2016 Jul 30;18:176. doi: 10.1186/s13075-016-1073-3. PMID 27473164
- [Background] Kosek E, Martinsen S, Gerdle B, Mannerkorpi K, Lofgren M, Bileviciute-Ljungar I, Fransson P, Schalling M, Ingvar M, Ernberg M, Jensen KB. The translocator protein gene is associated with symptom severity and cerebral pain processing in fibromyalgia. Brain Behav Immun. 2016 Nov;58:218-227. doi: 10.1016/j.bbi.2016.07.150. Epub 2016 Jul 20. PMID 27448744
- [Background] Ernberg M, Christidis N, Ghafouri B, Bileviciute-Ljungar I, Lofgren M, Larsson A, Palstam A, Bjersing J, Mannerkorpi K, Kosek E, Gerdle B. Effects of 15 weeks of resistance exercise on pro-inflammatory cytokine levels in the vastus lateralis muscle of patients with fibromyalgia. Arthritis Res Ther. 2016 Jun 13;18(1):137. doi: 10.1186/s13075-016-1041-y. PMID 27296860
- [Background] Palstam A, Larsson A, Lofgren M, Ernberg M, Bjersing J, Bileviciute-Ljungar I, Gerdle B, Kosek E, Mannerkorpi K. Decrease of fear avoidance beliefs following person-centered progressive resistance exercise contributes to reduced pain disability in women with fibromyalgia: secondary exploratory analyses from a randomized controlled trial. Arthritis Res Ther. 2016 May 21;18(1):116. doi: 10.1186/s13075-016-1007-0. PMID 27209068
- [Background] Christidis N, Ghafouri B, Larsson A, Palstam A, Mannerkorpi K, Bileviciute-Ljungar I, Lofgren M, Bjersing J, Kosek E, Gerdle B, Ernberg M. Comparison of the Levels of Pro-Inflammatory Cytokines Released in the Vastus Lateralis Muscle of Patients with Fibromyalgia and Healthy Controls during Contractions of the Quadriceps Muscle--A Microdialysis Study. PLoS One. 2015 Dec 1;10(12):e0143856. doi: 10.1371/journal.pone.0143856. eCollection 2015. PMID 26624891
- [Background] Flodin P, Martinsen S, Mannerkorpi K, Lofgren M, Bileviciute-Ljungar I, Kosek E, Fransson P. Normalization of aberrant resting state functional connectivity in fibromyalgia patients following a three month physical exercise therapy. Neuroimage Clin. 2015 Aug 18;9:134-9. doi: 10.1016/j.nicl.2015.08.004. eCollection 2015. PMID 26413476
- [Background] Larsson A, Palstam A, Lofgren M, Ernberg M, Bjersing J, Bileviciute-Ljungar I, Gerdle B, Kosek E, Mannerkorpi K. Resistance exercise improves muscle strength, health status and pain intensity in fibromyalgia--a randomized controlled trial. Arthritis Res Ther. 2015 Jun 18;17(1):161. doi: 10.1186/s13075-015-0679-1. PMID 26084281
- [Background] Martinsen S, Flodin P, Berrebi J, Lofgren M, Bileviciute-Ljungar I, Ingvar M, Fransson P, Kosek E. Fibromyalgia patients had normal distraction related pain inhibition but cognitive impairment reflected in caudate nucleus and hippocampus during the Stroop Color Word Test. PLoS One. 2014 Oct 2;9(9):e108637. doi: 10.1371/journal.pone.0108637. eCollection 2014. PMID 25275449
- [Background] Palstam A, Larsson A, Bjersing J, Lofgren M, Ernberg M, Bileviciute-Ljungar I, Ghafouri B, Sjors A, Larsson B, Gerdle B, Kosek E, Mannerkorpi K. Perceived exertion at work in women with fibromyalgia: explanatory factors and comparison with healthy women. J Rehabil Med. 2014 Sep;46(8):773-80. doi: 10.2340/16501977-1843. PMID 25074026
- [Background] Flodin P, Martinsen S, Lofgren M, Bileviciute-Ljungar I, Kosek E, Fransson P. Fibromyalgia is associated with decreased connectivity between pain- and sensorimotor brain areas. Brain Connect. 2014 Oct;4(8):587-94. doi: 10.1089/brain.2014.0274. Epub 2014 Aug 7. PMID 24998297
- [Derived] Wahlen K, Yan H, Welinder C, Ernberg M, Kosek E, Mannerkorpi K, Gerdle B, Ghafouri B. Proteomic Investigation in Plasma from Women with Fibromyalgia in Response to a 15-wk Resistance Exercise Intervention. Med Sci Sports Exerc. 2022 Feb 1;54(2):232-246. doi: 10.1249/MSS.0000000000002790. PMID 35029590
- [Derived] Sandstrom A, Ellerbrock I, Lofgren M, Altawil R, Bileviciute-Ljungar I, Lampa J, Kosek E. Distinct aberrations in cerebral pain processing differentiating patients with fibromyalgia from patients with rheumatoid arthritis. Pain. 2022 Mar 1;163(3):538-547. doi: 10.1097/j.pain.0000000000002387. PMID 34224497